CLINICAL TRIAL: NCT05619315
Title: Enamel Abrasion and Stain Removal Efficacy of Two Whitening Toothpastes
Brief Title: Enamel Abrasion and Stain Removal Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Metwally, bachelor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Charcoal based whitening
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Abrasion; Discoloration, Tooth
Keywords: abrasion; toothpaste; stain; whitening
MeSH Terms: conditions — Tooth Discoloration | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcoal -based whitening toothpaste. (Experimental): The labial surface of anterior teeth will be brushed by the circular brushing technique twice daily (morning and after 6 hours) for at least 1 minute using charcoal containing toothpaste. Soft bristles toothbrushes will provided to all patients. After 1 month, re-evaluation of the stains will be performed and the data will be recorded.
  Interventions: Other: Charcoal -based whitening toothpaste
- Calcium carbonate /perlite containing whitening toothpaste. (Active Comparator): The labial surface of anterior teeth will be brushed by the circular brushing technique twice daily (morning and after 6hours) for at least 1 minute using (calcium carbonate /perlite) containing toothpaste. Soft bristles toothbrushes will provided to all patients. After 1 month, re-evaluation of the stains will be performed and the data will be recorded.
  Interventions: Other: Calcium carbonate /perlite containing whitening toothpaste.

INTERVENTIONS:
Other: Charcoal -based whitening toothpaste — The labial surface of anterior teeth will be brushed by the circular brushing technique twice daily (morning and after 6 hours) for at least 1 minute using charcoal containing toothpaste. Soft bristles toothbrushes will provided to all patients. After 1 month, re-evaluation of the stains will be performed and the data will be recorded.
  Arms: Charcoal -based whitening toothpaste.
Other: Calcium carbonate /perlite containing whitening toothpaste. — The labial surface of anterior teeth will be brushed by the circular brushing technique twice daily (morning and after 6hours) for at least 1 minute using (calcium carbonate /perlite) containing toothpaste. Soft bristles toothbrushes will provided to all patients. After 1 month, re-evaluation of the stains will be performed and the data will be recorded.
  Arms: Calcium carbonate /perlite containing whitening toothpaste.

SUMMARY:
Enamel abrasion and stain removal efficacy of two whitening toothpastes

DETAILED DESCRIPTION:
Statement of the problem:

Access to in-office treatments is restricted to a lot of population. Therefore, there has been an interest in developing methods so that patients can remove stains and apply tooth whitening at home. Accordingly, toothpastes, due to their ease of use and low cost, have been used as vehicles for whitening agents as an alternative to home/office whitening.

Hydrogen peroxide is the most commonly used agent for whitening teeth, which is used in various concentrations according to various techniques at home and office. Bleaching of teeth in office is done at a high concentration of Hydrogen peroxide for a specified period of time. In addition to conventional whitening treatments, over-the-counter products, including gels, toothpastes, bleaching strips, mouthwashes, and pens with different Hydrogen peroxide levels, have been developed. In-office teeth whitening is one of the more costly forms of teeth whitening and the concentration of the bleaching element is higher, it is better monitored by a professional.

Whitening toothpaste is probably the one of the most affordable options for someone looking to whiten their teeth at home, which contain abrasive and chemical agents and have the ability to remove external stains from the tooth. The abrasiveness of toothpastes depends on the hardness, size, and shape of abrasive particles. Furthermore, factors such as the brushing technique, brushing pressure, toothbrush hardness, and the number of brush strokes affect tooth abrasion. Abrasive agents include silica, phosphates, carbonates, and bicarbonates Chemical agents present in whitening toothpastes are sodium citrate, phosphate salt, which react with chromogenic molecules of superficial dental stains and eliminate them from the tooth surface.

Whitening toothpastes include different active ingredients in their composition. It normally contain a higher amount of abrasives and detergents than do conventional toothpastes In this sense, it is important to point out that toothpastes with higher amounts of abrasives may produce increased surface roughness in dental tissues, or restorations, or even tooth sensitivity, especially if they are used routinely

Rationale:

Today, active charcoal is added to toothpastes which are marketed as charcoal toothpastes. The first report on the use of charcoal in oral and dental hygiene has been attributed to Hippocrates in ancient Greece. Charcoal is used as powder, soot, coal, and ash in different countries. Charcoal-based products are used in medical treatments, such as its use as an antidote for acute poisoning, drug overdose, skin infections, Charcoal is used legally for the coloring of food in China, Japan, and Korea to improve health.

Activated charcoal is produced as a natural method of the partial oxidation of various materials. High-porosity activated charcoal has the ability to exchange ion in the mouth through nanopores and can attach to tooth enamel and remove tooth-coloring agents (because of its capacity of adsorbing pigments, chromophores, and stains from the tooth surface). The application of this product has been suggested to eliminate some dental coloring agents. Charcoal can help tooth whitening through tooth abrasion.

ELIGIBILITY:
Inclusion Criteria:

In vivo:

* Patients inclusion:

  1. Adult male and female patients ≥18 years.
  2. Good oral and general health and oral hygiene have at least eight natural anterior teeth (incisors and canines) assessable for extrinsic stain and be available for all study appointments.

Tooth inclusion:

Vital anterior maxillary and mandibular teeth free of caries or restorations, no cervical lesions and no periodontal disease.

In vitro:

Teeth inclusion criteria:

1. Intact, free of caries or restorations.
2. No cervical lesions .

Exclusion Criteria:

In vivo:

Patients exclusion:

1. Uncooperative behavior.
2. Patients allergic to tooth paste material.
3. Patient with history of medical disease, drug therapies or any other serious relevant problem.
4. Pregnant or breastfeeding women.
5. Patients with fixed orthodontic appliances
6. Patients who had professional tooth whitening, within the last six months.
7. Patients who had significant amounts of calculus on facial surfaces of the incisors/canines.
8. Patients who had undergone professional periodontal treatment within the previous six months or used mouth rinses for the treatment/ control of a periodontal condition.
9. Patients who had advanced periodontal disease on anterior teeth.
10. Xerostomic patients.
11. Patients who used medications which could affect saliva flow or cause staining.
12. Patients who had undergone dental prophylaxis within 8 weeks of screening.
13. Patients who used minocycline or doxycycline within 30 days of screening or between screening and baseline

Tooth exclusion:

1. Intrinsically Discolored teeth caused by tetracycline, fluorosis, hypocalcification hyperplasia, endodontic treatment (or requiring endodontic treatment).
2. Restorations in anterior teeth, parafunctional habits or tooth sensitivity.
3. Non- vital teeth

In vitro:

Teeth exclusion criteria:

1. Intrinsically Discolored teeth caused by tetracycline, fluorosis, hyperplasia, endodontic treatment .
2. Restorations in teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Stain score | T0: Baseline
  mcpherson modification of the stain index and area x intensity
Stain score | T1: 4 weeks
  mcpherson modification of the stain index and area x intensity

SECONDARY OUTCOMES:
Surface roughness | T0: Baseline
  Atomic Force Microscopy
Surface roughness | T1: 3 minutes equivalent to 2 times a day for one month.
  Atomic Force Microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Iman Ibrahim El Sayad, prof, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghassemi A, Hooper W, Vorwerk L, Domke T, DeSciscio P, Nathoo S. Effectiveness of a new dentifrice with baking soda and peroxide in removing extrinsic stain and whitening teeth. J Clin Dent. 2012;23(3):86-91. PMID 23210419
- [Background] Watts A, Addy M. Tooth discolouration and staining: a review of the literature. Br Dent J. 2001 Mar 24;190(6):309-16. doi: 10.1038/sj.bdj.4800959. PMID 11325156
- [Background] Lima DA, Silva AL, Aguiar FH, Liporoni PC, Munin E, Ambrosano GM, Lovadino JR. In vitro assessment of the effectiveness of whitening dentifrices for the removal of extrinsic tooth stains. Braz Oral Res. 2008 Apr-Jun;22(2):106-11. doi: 10.1590/s1806-83242008000200003. PMID 18622478
- [Background] Kalyana P, Shashidhar A, Meghashyam B, Sreevidya KR, Sweta S. Stain removal efficacy of a novel dentifrice containing papain and Bromelain extracts--an in vitro study. Int J Dent Hyg. 2011 Aug;9(3):229-33. doi: 10.1111/j.1601-5037.2010.00473.x. Epub 2010 Jul 1. PMID 21356017
- [Background] Collins LZ, Naeeni M, Schafer F, Brignoli C, Schiavi A, Roberts J, Colgan P. The effect of a calcium carbonate/perlite toothpaste on the removal of extrinsic tooth stain in two weeks. Int Dent J. 2005;55(3 Suppl 1):179-82. doi: 10.1111/j.1875-595x.2005.tb00056.x. PMID 16004250
- [Background] Patil PA, Ankola AV, Hebbal MI, Patil AC. Comparison of effectiveness of abrasive and enzymatic action of whitening toothpastes in removal of extrinsic stains - a clinical trial. Int J Dent Hyg. 2015 Feb;13(1):25-9. doi: 10.1111/idh.12090. Epub 2014 Jul 21. PMID 25046241
- [Background] Zafar MS, Ahmed N. Nanomechanical characterization of exfoliated and retained deciduous incisors. Technol Health Care. 2014;22(6):785-93. doi: 10.3233/THC-140852. PMID 25134963
- [Background] Litonjua LA, Andreana S, Bush PJ, Tobias TS, Cohen RE. Noncarious cervical lesions and abfractions: a re-evaluation. J Am Dent Assoc. 2003 Jul;134(7):845-50. doi: 10.14219/jada.archive.2003.0282. PMID 12892441
- [Background] Johannsen G, Tellefsen G, Johannsen A, Liljeborg A. The importance of measuring toothpaste abrasivity in both a quantitative and qualitative way. Acta Odontol Scand. 2013 May-Jul;71(3-4):508-17. doi: 10.3109/00016357.2012.696693. Epub 2012 Jul 2. PMID 22746180
- [Background] Carey CM. Tooth whitening: what we now know. J Evid Based Dent Pract. 2014 Jun;14 Suppl:70-6. doi: 10.1016/j.jebdp.2014.02.006. Epub 2014 Feb 13. PMID 24929591
- [Background] Ozkan P, Kansu G, Ozak ST, Kurtulmus-Yilmaz S, Kansu P. Effect of bleaching agents and whitening dentifrices on the surface roughness of human teeth enamel. Acta Odontol Scand. 2013 May-Jul;71(3-4):488-97. doi: 10.3109/00016357.2012.696691. Epub 2012 Jul 2. PMID 22747485
- [Background] Barbieri GM, Mota EG, Rodrigues-Junior SA, Burnett LH Jr. Effect of whitening dentifrices on the surface roughness of commercial composites. J Esthet Restor Dent. 2011 Oct;23(5):338-45. doi: 10.1111/j.1708-8240.2011.00426.x. Epub 2011 May 9. PMID 21977958
- [Background] Gerlach RW, Barker ML, Tucker HL. Clinical response of three whitening products having different peroxide delivery: comparison of tray, paint-on gel, and dentifrice. J Clin Dent. 2004;15(4):112-7. PMID 15794456
- [Background] Joiner A. Review of the extrinsic stain removal and enamel/dentine abrasion by a calcium carbonate and perlite containing whitening toothpaste. Int Dent J. 2006 Aug;56(4):175-80. doi: 10.1111/j.1875-595x.2006.tb00091.x. PMID 16972390
- [Background] Brooks JK, Bashirelahi N, Reynolds MA. Charcoal and charcoal-based dentifrices: A literature review. J Am Dent Assoc. 2017 Sep;148(9):661-670. doi: 10.1016/j.adaj.2017.05.001. Epub 2017 Jun 7. PMID 28599961
- [Background] Pintado-Palomino K, Vasconcelos CV, Silva RJ, Fressatti AL, Motta BJ, Pires-DE-Souza FC, Tirapelli C. Effect of whitening dentifrices: a double-blind randomized controlled trial. Braz Oral Res. 2016 Oct 10;30(1):e82. doi: 10.1590/1807-3107BOR-2016.vol30.0082. PMID 27737352
- [Background] Joiner A. Whitening toothpastes: a review of the literature. J Dent. 2010;38 Suppl 2:e17-24. doi: 10.1016/j.jdent.2010.05.017. Epub 2010 May 24. PMID 20562012
- [Background] Wulknitz P. Cleaning power and abrasivity of European toothpastes. Adv Dent Res. 1997 Nov;11(4):576-9. doi: 10.1177/08959374970110042701. PMID 9470519
- [Background] Joiner A, Philpotts CJ, Alonso C, Ashcroft AT, Sygrove NJ. A novel optical approach to achieving tooth whitening. J Dent. 2008;36 Suppl 1:S8-14. doi: 10.1016/j.jdent.2008.02.005. PMID 18646364
- [Background] Macpherson LM, Stephen KW, Joiner A, Schafer F, Huntington E. Comparison of a conventional and modified tooth stain index. J Clin Periodontol. 2000 Nov;27(11):854-9. doi: 10.1034/j.1600-051x.2000.027011854.x. PMID 11073329
- [Background] Black MA, Bayne SC, Peterson CA. Effect of power toothbrushing on simulated wear of dental cement margins. J Dent Hyg. 2007 Fall;81(4):79. Epub 2007 Oct 1. PMID 18173893
- [Background] Hattab FN, Qudeimat MA, al-Rimawi HS. Dental discoloration: an overview. J Esthet Dent. 1999;11(6):291-310. doi: 10.1111/j.1708-8240.1999.tb00413.x. PMID 10825865